CLINICAL TRIAL: NCT01021943
Title: The Role of Spironolactone in Prevention of Calcineurin Inhibitor Toxicity in Kidney Transplant Recipients
Brief Title: Spironolactone and Prevention of Calcineurin Inhibitor Toxicity in Kidney Transplant Recipients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Magdalena Madero, Chief Nephrology Division, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT-26
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Transplant
Keywords: calcineurin inhibitors; fibrosis; spironolactone; Focus of the study is to assess if aldosterone blockade has an effect on interstitial fibrosis amongst kidney transplant recipients
MeSH Terms: conditions — Fibrosis | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Half of the subjects will be assigned to receive either spironolactone or placebo for 6 months
  Interventions: Drug: Placebo
- spironolactone (Active Comparator): Half of the subjects will be randomized to receive spironolactone for 6 months
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone — Half of the subjects will be assigned to receive 25 mg of spironolactone for 6 months
  Arms: spironolactone
Drug: Placebo — Half of the subjects will be assigned to receive placebo for 6 months
  Arms: Placebo

SUMMARY:
The main objective of this study is to assess the effect of spironolactone on interstitial fibrosis in kidney transplant recipients receiving calcineurin inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Kidney Failure
* Age > 18
* Kidney transplant recipients

Exclusion Criteria:

* Patients taking angiotensin receptor blockers or inhibitors of the angiotensin reconverting enzyme
* Kidney transplant performed more than one month from enrollment in the study
* Hyperkalemia (K> 5.5 meqL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-11

PRIMARY OUTCOMES:
Interstitial fibrosis in kidney transplant biopsies (time zero biopsy and at 6 months post intervention) | 2 years

SECONDARY OUTCOMES:
allograft function and proteinuria | 2 years
Fibrosis markers in kidney biopsies such as TGF-B | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional Nutricion Salvador Zubiran, México, Mexico